CLINICAL TRIAL: NCT01449825
Title: Postmarketing Hepatic Monitoring for Pazopanib Using Observational Databases
Brief Title: Hepatic Monitoring for Pazopanib
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114430; WEUKSTV4601 (Other: GSK)
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: hepatic safety; prescriber compliance; pazopanib; epidemiology
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prescriber compliance group: Adult (18+ years) new users of pazopanib with an indication of RCC evaluated for prescriber compliance
  Interventions: Drug: Pazopanib use
- Incidence of liver chemistry test (LCT) elevation group: Adult (18+ years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib in monotherapy who have a baseline LCT evaluated for LCT elevations
  Interventions: Drug: Pazopanib use; Drug: Use of sunitinib, bevacizumab, or sorafenib
- Incidence of drug induced liver injury (DILI) cases group: Adult (18+ years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib with RCC (as defined by ICD-9 codes) longitudinally followed up in order to capture occurrences of LCT elevations consistent with Hy's Law to evaluate for drug-induced liver injury
  Interventions: Drug: Pazopanib use; Drug: Use of sunitinib, bevacizumab, or sorafenib
- Incidence of cases of ALF group: Adult (18+ years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib with RCC (as defined by ICD-9 codes) longitudinally followed up in order to capture occurrences of ICD-9 codes indicative of possible ALF to evaluate for drug-induced liver injury
  Interventions: Drug: Pazopanib use; Drug: Use of sunitinib, bevacizumab, or sorafenib

INTERVENTIONS:
Drug: Pazopanib use — Treatment with pazopanib
Drug: Use of sunitinib, bevacizumab, or sorafenib — Treatment with any of the three other marketed anti-VEGF drugs: sunitinib, bevacizumab, and sorafenib
  Groups: Incidence of cases of ALF group; Incidence of drug induced liver injury (DILI) cases group; Incidence of liver chemistry test (LCT) elevation group

SUMMARY:
Pazopanib is approved by the FDA and EMA as targeted therapy for the indication of advanced renal cell carcinoma (RCC). Hepatic safety events were observed in the pazopanib pivotal clinical trial and the U.S. pazopanib label information contains a 'black box warning' regarding hepatotoxicity. These clinical observations have prompted GSK to undertake a proactive pharmacovigilance strategy focused on hepatic safety that goes beyond spontaneous reporting of adverse events.

The goals of the study are to assess prescriber compliance with pazopanib label guidelines for liver monitoring among patients with RCC, as well as to quantify and characterize the hepatic safety profile of the product in real-world clinical practice compared to other anti-vascular endothelial growth factor (anti-VEGF) drugs. As part of regulatory commitments, GSK will conduct parallel epidemiologic analyses in different patient populations as represented in multiple databases of electronic medical records. To enhance accrual of data, GSK will conduct this safety surveillance program simultaneously across datasets in order to detect and characterize all cases of liver enzyme elevations in diverse populations of patients receiving pazopanib. Two additional goals of this study are to evaluate the incidence of cases of combinations of liver enzyme elevations indicative of Hy's Law and drug-induced acute liver failure among users of pazopanib compared to users of other anti-VEGF drugs. This research effort will be coordinated by an external coordinating center.

An epidemiologic cohort study design, nested in several databases of electronic medical information, will be employed for the research questions. Following the availability of pazopanib in the relevant medical care system, the study will collect retrospective data at regular intervals over the course of four years among persons exposed to pazopanib and other anti-VEGF agents. Each patient will be characterized based on additional available information in the database (e.g., demographics, concomitant medications). Elevations in liver enzymes will be identified through laboratory data captured in these databases. Potential Hy's Law and acute liver failure cases will be identified through established screening criteria, and screen-positive cases will be reviewed by an adjudication committee of hepatologists for final determination of drug-associated causality.

ELIGIBILITY:
Inclusion Criteria:

* In the prescriber compliance analysis, all adult (18+ years) new users of pazopanib with an indication of RCC will be eligible for the analysis.
* In the liver enzyme elevation analysis, all adult (18+ years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib in monotherapy for any cancer type who have a baseline liver enzyme value will be eligible for the analysis.
* In the drug-induced liver injury analyses, all adult (18+ years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib with RCC (as defined by ICD-9 codes) will be longitudinally followed up in order to capture occurrences of liver enzyme elevations consistent with Hy's Law and ICD-9 codes indicative of possible ALF to evaluate for drug-induced liver injury.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult (18+years) new users of pazopanib, sunitinib, bevacizumab, and sorafenib.
  Two U.S. healthcare databases and one Dutch-linked medical registry system will contribute de-identified and anonymised data from electronic medical records to the surveillance program.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prescriber compliance with pazopanib label guidelines for liver monitoring | Over four years of treatment with pazopanib
  Prescriber compliance with pazopanib label guidelines for liver monitoring
Incidence of liver enzyme elevations including combination liver enzyme elevations suggestive of Hy's Law | Over four years of treatment with pazopanib
  Incidence of liver enzyme elevations including combination liver enzyme elevations suggestive of Hy's Law
Incidence of acute liver failure (ALF) | Over four years of treatment with pazopanib
  Incidence of ALF

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline